CLINICAL TRIAL: NCT02978599
Title: Double Blind, Two Dose, Cross-over Clinical Trial of the Positive Allosteric Modulator at the alpha7 Nicotinic Cholinergic Receptor AVL-3288 in Schizophrenia Patients
Brief Title: Clinical Trial of AVL-3288 in Schizophrenia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joshua Kantrowitz, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 7370; U01MH094247-01 (NIH)
Record Dates: First submitted 2016-11-17; First posted 2016-12-01 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — AVL3288

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AVL-3288 10 mg (Experimental): AVL-3288 10 mg daily for 5 days
  Interventions: Drug: AVL-3288
- AVL-3288 30 mg (Experimental): AVL-3288 30 mg daily for 5 days
  Interventions: Drug: AVL-3288
- Placebo (Placebo Comparator): Placebo daily for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVL-3288 — daily for 5 days
  Other Names: Anvylic-3288
  Arms: AVL-3288 10 mg; AVL-3288 30 mg
Drug: Placebo — daily for 5 days
  Arms: Placebo

SUMMARY:
Single-center, outpatient, randomized, double-blind, placebo-controlled, 3-treatment-phase, cross-over study to evaluate the safety, tolerability and efficacy of two oral doses of AVL-3288 each compared to placebo, in patients with schizophrenia.

DETAILED DESCRIPTION:
This study will be in 24 non-smoking outpatients with schizophrenia or schizoaffective disorder. Subjects will complete three treatment phases, each involving 5 straight days of taking AVL-3288 (10 mg or 30 mg study drug or placebo) followed by a 16 day washout period in which subjects do not take the study drug to ensure that the drug is completed eliminated from the body before the next phase.

ELIGIBILITY:
Inclusion Criteria:

* DSM-V diagnosis of schizophrenia or schizoaffective disorder
* RBANS Total Scale Score >62
* Willing to provide informed consent
* Medically stable for study participation
* Taking an antipsychotic medication other than clozapine at a stable dose for at least 4 weeks
* Judged clinically not to be at significant suicide or violence risk

Exclusion Criteria:

* Substance abuse (excluding nicotine) within last 90 days
* ECG abnormality that is clinically significant
* Current clozapine use
* Participation in a study of investigational medication/device within 4 weeks
* Pregnancy, lactation, or lack of use of effective birth control
* Active tobacco use
* Presence or positive history of significant medical or neurological illness, including cardiac illness, WBC <3500/mm3, absolute neutrophil count <1500/mm3, ALT or AST values >1.5 times upper limit of normal. Hemoglobin less than 130 g/L (13 g/dL) in males or 120 g/L (12 g/dL) in females or known HIV +
* Contraindication to MRI scanning, including metal implants or claustrophobia
* Medicinal patch, unless removed

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11; Primary Completion 2018-10-26 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Total Scale Score | End of each 5-day treatment phase
  Compare effect of active drug (AVL-3288) to placebo on RBANS total score

SECONDARY OUTCOMES:
RBANS index T-score subscales | End of each 5-day treatment phase
  Compare effect of active drug (AVL-3288) to placebo on RBANS index T-score subscales
Brief Psychiatric Rating Scale (BPRS) Total score | End of each 5-day treatment phase
  Compare effect of active drug (AVL-3288) to placebo on BPRS Total Score.
Calgary Depression Rating Scale (CDRS) Total score | End of each 5-day treatment phase
  Compare effect of active drug (AVL-3288) to placebo on CDRS Total Score.
Scale for the Assessment of Negative Symptoms (SANS) Total score | End of each 5-day treatment phase
  Compare effect of active drug (AVL-3288) to placebo on SANS Total score
P50 suppression measured by electroencephalographic (EEG) | End of each 5-day treatment phase
  Compare P50 suppression measured by EEG between active drug (AVL-3288) and placebo
Intensity of hippocampal BOLD fMRI signal during MRI scan | end of each 5-day treatment phase
  Compare intensity of Hippocampal BOLD signal between active drug (AVL-3288) and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Lieberman, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes